CLINICAL TRIAL: NCT05237999
Title: KopOpOuders-PTSD: Randomized Controlled Trial of A Preventive Blended Care Parenting Intervention for Parents With PTSD
Brief Title: Effectiveness of a Blended Care Parenting Intervention for Parents With PTSD (KopOpOuders-PTSD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arkin (Industry)
Collaborators: Sinai Centrum (Unknown); Trimbos Institute (Unknown); Arkin Jeugd en Gezin Preventie (Unknown); Utrecht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOO-PTSS
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Post-traumatic Stress Disorder
Keywords: post-traumatic stress disorder; parenting; children of parents with mental illness (COPMI); social support
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial comparing KopOpOuders-PTSD to control (no intervention). In the intervention group, participants complete 8 sessions over 9 weeks (5 individual online self-help modules, 3 in-person sessions with a prevention professional) of KopOpOuders-PTSD. In the control group, participants do not receive an intervention (but do get access to the online self-help modules after their participation). In both conditions, PTSD treatment (and other therapies if applicable) continue as normal during and after participation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments will be performed by allocation-blind assessors. The randomization procedure is carried out by a research assistant not involved in assessments, and outcomes are not visible for assessors. Participants are reminded immediately at each contact with an assessor that they are not allowed to discuss whether or not they were in the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: KopOpOuders-PTSD (Experimental): KopOpOuders-PTSD is a blended care (i.e., partially online and partially in person) intervention that addresses the enhancing of protective factors within the family setting (reducing negative parental self-perceptions; parent-child interaction quality, social support, child adaptive functioning/coping, and child understanding of the parent's illness) from a combination of transdiagnostic and PTSD-specific perspectives. It consists of 8 sessions (5 online self-help modules, 3 in-person sessions with a professional) to be completed in a maximum period of 9 weeks.
  Interventions: Behavioral: KopOpOuders-PTSD
- Control: No intervention (No Intervention): The control group receives no parenting intervention during their participation.

INTERVENTIONS:
Behavioral: KopOpOuders-PTSD — See arm description
  Other Names: KopOpOuders for PTSD
  Arms: Intervention: KopOpOuders-PTSD

SUMMARY:
KopOpOuders-PTSD is a new preventive blended care intervention for parents with PTSD. The purpose of this study is to evaluate its effectiveness in improving parenting and preventing child mental health problems.

DETAILED DESCRIPTION:
Rationale: Children of parents with post-traumatic stress disorder (PTSD) are at increased risk of mental health problems, such as depression, anxiety and hyperactivity. They are also more likely than children of healthy parents to be exposed to potential trauma, especially in the family setting (e.g., child maltreatment). Parents with PTSD often experience difficulties in their parenting role (e.g., deficits in effective parenting, sense of parenting incompetence, lack of social support). Research in other mental disorders shows that preventively supporting parents with mental illness in their parenting role decreases mental health problems in children. As of yet, no preventive intervention specifically aimed at parents with PTSD exist. We have therefore adapted an existing preventive online course for parents with mental illness, 'KopOpOuders zelfhulp', into a blended care intervention for parents with PTSD: 'KopOpOuders-PTSD'. This intervention was developed in co-creation with parents with PTSD and their partners.

Objective: Main objective: to test the effectiveness of KopOpOuders-PTSD on macro- and micro-level parenting behavior. Secondary objectives: to test the effectiveness of KopOpOuders-PTSD on perceived parenting competence, parents' social support, and child mental health; to test whether intervention effects are moderated by baseline PTSD symptoms.

Study design: The study uses a single-blind randomized controlled trial design with three measurement points (pretest, posttest, and follow-up). Data are collected through self-report questionnaires (macro-level) and ecological momentary assessment (EMA; micro-level) using a smartphone app.

Study population: 142 adults (71 per condition) receiving PTSD treatment at Arkin (departments Sinai Centrum, NPI, Jellinek, Arkin Basis GGZ), who have parenting responsibilities for one or more children aged 4-17.

Intervention (if applicable): The intervention group receives KopOpOuders-PTSD, consisting of 5 online modules and 3 face-to-face sessions, in addition to treatment as usual. The control group does not receive intervention apart from treatment as usual, but can access the online modules of KopOpOuders-PTSD after participation.

Main study parameters/endpoints: Main study parameters are mean level change from pretest to posttest in parenting behavior at the macro- and micro-level.

ELIGIBILITY:
Inclusion criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Has current DSM-5 diagnosis of PTSD;
* Is receiving PTSD treatment of at least three sessions at one of the following Arkin departments: Sinai Centrum, Jellinek, Punt P, NPI, or Arkin BasisGGZ;
* Has parenting responsibilities for at least one child aged 4-17 (biological or legal relationship not required).

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Has urgent care needs or (imminent) crisis (e.g. current psychosis, substance detoxification, active suicidality);
* Is not in contact with children (e.g. due to out of home placement);
* Is receiving another form of parenting intervention during the participation period;
* Severe psychological problems or intellectual disability (IQ < 50) are present in children (diagnosis of oppositional-defiant disorder, conduct disorder, psychotic spectrum disorder or personality disorder);
* Inability to participate in the intervention and/or assessments (e.g., because of intellectual disability (IQ < 75), illiteracy, or insufficient mastery of the Dutch language).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Alabama Parenting Questionnaire (APQ) | 2 months
  Parenting skills are measured using the caregiver-report version of the Alabama Parenting Questionnaire (APQ; Frick, 1991). The APQ is a 42-item questionnaire with five subscales: positive involvement with children, supervision/monitoring, use of positive discipline techniques, consistency in discipline techniques, and use of corporal punishment. Responses are scored on a five-point Likert scale ranging from 'never' (1) to 'always' (5). APQ total scores range from 42 to 210. We will recode items so that higher scores reflect more positive parenting. The total score will be used for the main analysis and we will perform additional analyses on the separate subscales. We will use the Dutch translation of the APQ (Van Lier & Crijnen, 1999).
Short Parenting Scale for EMA (SPS-EMA) | 5 hours
  Parenting behavior is assessed three times a day during two weeks (at baseline and posttest) with an app for ecological momentary assessment (EMA) using eight adapted items from the Parenting Behavior Inventory (PBI; Lovejoy et al., 1999). For this study, we have selected eight items from the PBI, of which four from each subscale (hostile/coercive and supportive/engaged). The wording of these items has been changed slightly to fit with the EMA format (e.g., 'I say mean things to my child that could make him/her feel bad' becomes 'Since the last notification… I have said mean things to my child that could make him/her feel bad'). We have also changed the response scale from seven- to three-point Likert scale: 'Not true' (1), 'Somewhat true' (2), 'Certainly true' (3). We will analyze the total score of the two subscales combined which ranges from 8-24. For this study, we will call this questionnaire the 'Short Parenting Scale for EMA' (SPS-EMA).

SECONDARY OUTCOMES:
Parenting Sense of Competence Scale (PSOCS) | 2 months
  Perceived parenting competence is measured using the Parenting Sense of Competence Scale (PSOCS; Johnston & Mash, 1989). The PSOCS is a 17-item questionnaire comprising two subscales: satisfaction and efficacy. We will use the total score for the main analysis and perform additional analyses on the two subscales. Items are posed as statements (e.g., 'Being a parent makes me tense and anxious'), which are scored for agreement on a six-point Likert scale ranging from 'strongly disagree' (1) to 'strongly agree' (6). PSOCS total scores range from 17 to 102. We will use the Dutch translation of the PSOCS.
Interpersonal Social Support Evaluation List - 12 | 2 months
  Parent social support is measured using the abbreviated version of the Interpersonal Social Support Evaluation List (ISEL-12 (72)). The ISEL-12 has 12 items comprising three subscales: appraisal support, belonging support, and tangible support. We will use the total score for our main analysis (research question 4). Items are rated on a four-point scale ranging from 'Definitely false' (1) to 'Definitely true' (4). ISEL-12 total scores range from 12-48, and will be coded so that higher scores indicate more support. The ISEL-12 total score has good psychometric properties (Cohen et al., 1985). We translated the ISEL-12 to Dutch using the back-translation method. We also added two self-made items reflecting aspects of social support we were interested in in light of our intervention: having someone to look after your children (tangible support) and having someone to talk to about worries about your child (appraisal support). These will be analyzed descriptively.
Strengths and Difficulties Questionnaire - Parent Report (SDQ-P) | 2 months
  Child overall psychological problems are measured using parent-report on the Strengths and Difficulties Questionnaire-Parent Report (SDQ-P; Goodman, 1997). The SDQ-P. The SDQ-P comprises five subscales with five items each: hyperactivity/attention deficit, emotional problems, behavioral problems, peer relationship problems, and prosocial behavior. We will use the 'general difficulties' score as our analysis outcome, which aggregates all subscales excluding prosocial behavior (thus comprising 20 items). We will perform additional analyses on the separate subscales. Items are scored on a three-point Likert scale ranging from 'Not true' (0) to 'Certainly true' (2). The 'general difficulties' score ranges from 0-40. We will use the Dutch translation of the SDQ-P (van Widenfelt et al., 2003).
Child and Adolescent Trauma Screener-Caregiver Report (CATS-C) | 2 weeks
  Child PTSD symptoms are measured using parent-report on the Child and Adolescent Trauma Screener-Caregiver Report (CATS-C; Sachser et al., 2017; Dutch translation: Kooij & Lindauer, 2022). The CATS-C starts with 15 yes/no items about child exposure to DSM-5 A-criterion traumatic events. If the parent reports their child has been exposed to at least one of these events, the questionnaire continues with 16 (age 3-6) or 20 (age 7-17) items about PTSD symptoms. Data on PTSD symptoms are thus only collected if the child has experienced at least one A-criterion traumatic event. PTSD symptom items are rated on a four-point Likert scale ranging from 'Never' (0) to 'Almost always' (3). Interference with life domains is assessd with five yes/no items. We will analyze the total symptom score (range: 0-48 for age 3-6; 0-60 for age 7-17). We will perform additional analyses on the separate subscales. Scores on trauma exposure items will be reported descriptively.

OTHER OUTCOMES:
PTSD Checklist for DSM-5 | 1 month
  PTSD symptoms are measured at baseline using the PTSD Checklist for DSM-5 (PCL-5; Blevins et al., 2015). The PCL-5 comprises 20 items describing PTSD symptoms rated on a five-point Likert scale ranging from 'Not at all' (0) to 'Extremely' (4). The PCL-5 comprises four subscales corresponding to DSM-5 PTSD symptom clusters (intrusion, avoidance, negative alterations in mood and cognitions, and hyperarousal). We will use the PCL-5 total score (ranging from 0-80) as a moderator variable. We will use the Dutch translation of the PCL-5 (Boeschoten et al., 2014).
Life Events Questionnaire for DSM-5 (LEC-5) | Lifetime
  Trauma exposure is measured at baseline using the Life Events Questionnaire for DSM-5 (LEC-5; Weathers et al., 2013). The LEC-5 comprises 17 items which describe DSM-5 A-criterion traumatic events (e.g., 'Fire or explosion'). Participants note for each event on a scale with 6 options whether they were directly or indirectly (i.e., as a witness, learning about it happening to someone close to them, or as part of their job) exposed to it. In case of multiple trauma exposures, the participant is asked to indicate which event bothers them the most. This event is called the 'index trauma' and will be used to determine trauma type in this study. The Dutch translation of the LEC-5 is used (Boeschoten et al., 2014).
Outcome Questionnaire-45 (OQ-45) | 1 week
  General psychosocial functioning is measured as part of the ROM at Arkin using the Outcome Questionnaire-45 (OQ-45; Lambert et al., 1996). We will use the closest ROM measurement before baseline. The OQ-45 comprises 45 items, divided into three subscales: symptom distress (25 items, measures symptoms of depression, anxiety and substance abuse), interpersonal relations (11 items, measures relational functioning) and social role (9 items, measures functioning in school, work and/or leisure). Items are scored on a 5-point Likert scale ranging from 'Never' (0) to 'Always' (4). We will descriptively report the OQ-45 total score, which ranges from 0-180.
Demographic information | Lifetime
  To provide information on the demographic background of the sample, participants complete a short demographic questionnaire (DQ) at baseline with items about themselves and their children.
Intervention adherence and satisfaction | 10 weeks
  For participants in the intervention condition, results on intervention adherence (completion of online modules; attendance of face-to-face sessions; and use of PTSD-specific content in the online library) will be reported descriptively. Furthermore, intervention group participants complete a short satisfaction questionnaire (SQ) at posttest. The SQ contains closed-ended and open-ended questions on aspects of the intervention, and invites participants to provide suggestions for improvement. Results will be reported descriptively in the publication of the current study and will be used for future improvement of the intervention.
Short Form PTSD Checklist for DSM-5 (SF-PCL-5) | 5 hours
  PTSD symptoms are assessed in the EMA app using a short-form version of the PTSD Checklist for DSM-5 (PCL-5) with one item for each of the four symptom clusters (SF-PCL-5; Zuromski et al., 2019). Each item is rated for past-month frequency on a five-point Likert scale ranging from 'Not at all' (0) to 'Extremely' (4). The instruction of the SF-PCL-5 will be changed to fit with the EMA format. That is, participants are asked to report on their symptoms during the current part of the day (morning/afternoon/evening). Scores range from 0-16.
Sleep Quality Rating | 1 day
  Sleep quality will only be assessed in the morning EMA assessments, using a single item ('How well did you sleep last night?') answered on a 10-point scale.
Situational Context | 5 hours
  To assess the situational context, each EMA questionnaire starts with two situation items (Where are you; Who are you with), answered using multiple choice.
Distress Rating | 5 hours
  To assess current levels of distress, each EMA questionnaire contains a single item ('How much distress are you currently feeling?'), answered on a 10-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Thomaes, Principal Investigator — Sinai Centrum
Locations (1):
- Sinai Centrum, Amstelveen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, metadata will be made available. Anonymized IPD can be requested by submitting a data request form to the investigators. IPD will only be shared for those participants who provided informed consent for this in advance.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Anticipated in 2025, for at least 15 years.
Access Criteria: Data request form

REFERENCES:
- [Background] Bowers ME, Yehuda R. Intergenerational Transmission of Stress in Humans. Neuropsychopharmacology. 2016 Jan;41(1):232-44. doi: 10.1038/npp.2015.247. Epub 2015 Aug 17. PMID 26279078
- [Background] Chesmore AA, Piehler TF, Gewirtz AH. PTSD as a moderator of a parenting intervention for military families. J Fam Psychol. 2018 Feb;32(1):123-133. doi: 10.1037/fam0000366. Epub 2017 Dec 28. PMID 29283597
- [Background] Christie H, Hamilton-Giachritsis C, Alves-Costa F, Tomlinson M, Halligan SL. The impact of parental posttraumatic stress disorder on parenting: a systematic review. Eur J Psychotraumatol. 2019 Jan 14;10(1):1550345. doi: 10.1080/20008198.2018.1550345. eCollection 2019. PMID 30693071
- [Background] Chun CA. The Expression of Posttraumatic Stress Symptoms in Daily Life: A Review of Experience Sampling Methodology and Daily Diary Studies. Journal of Psychopathology and Behavioral Assessment. 2016; 38(3): 406-420.
- [Background] Hosman CMH, van Doesum KTM, van Santvoort F. Prevention of emotional problems and psychiatric risks in children of parents with a mental illness in the Netherlands: I. The scientific basis to a comprehensive approach. Australian E-Journal for the Advancement of Mental Health. 2006; 8(3): 250-263.
- [Background] Jones TL, Prinz RJ. Potential roles of parental self-efficacy in parent and child adjustment: a review. Clin Psychol Rev. 2005 May;25(3):341-63. doi: 10.1016/j.cpr.2004.12.004. PMID 15792853
- [Background] Lambert JE, Holzer J, Hasbun A. Association between parents' PTSD severity and children's psychological distress: a meta-analysis. J Trauma Stress. 2014 Feb;27(1):9-17. doi: 10.1002/jts.21891. Epub 2014 Jan 24. PMID 24464491
- [Background] Leen-Feldner EW, Feldner MT, Knapp A, Bunaciu L, Blumenthal H, Amstadter AB. Offspring psychological and biological correlates of parental posttraumatic stress: review of the literature and research agenda. Clin Psychol Rev. 2013 Dec;33(8):1106-33. doi: 10.1016/j.cpr.2013.09.001. Epub 2013 Sep 12. PMID 24100080
- [Background] Montgomery E, Just-Ostergaard E, Jervelund SS. Transmitting trauma: a systematic review of the risk of child abuse perpetrated by parents exposed to traumatic events. Int J Public Health. 2019 Mar;64(2):241-251. doi: 10.1007/s00038-018-1185-4. Epub 2018 Dec 1. PMID 30506365
- [Background] Siegenthaler E, Munder T, Egger M. Effect of preventive interventions in mentally ill parents on the mental health of the offspring: systematic review and meta-analysis. J Am Acad Child Adolesc Psychiatry. 2012 Jan;51(1):8-17.e8. doi: 10.1016/j.jaac.2011.10.018. Epub 2011 Dec 3. PMID 22176935
- [Background] Thanhauser M, Lemmer G, de Girolamo G, Christiansen H. Do preventive interventions for children of mentally ill parents work? Results of a systematic review and meta-analysis. Curr Opin Psychiatry. 2017 Jul;30(4):283-299. doi: 10.1097/YCO.0000000000000342. PMID 28505032
- [Background] Thomas JC, Letourneau N, Campbell TS, Giesbrecht GF; Apron Study Team. Social buffering of the maternal and infant HPA axes: Mediation and moderation in the intergenerational transmission of adverse childhood experiences. Dev Psychopathol. 2018 Aug;30(3):921-939. doi: 10.1017/S0954579418000512. PMID 30068422
- [Background] van Doesum, K. T. Databank effectieve jeugdinterventies: Beschrijving 'KopOpOuders'. Nederlands Jeugdinstituut. 2020.
- [Background] van Ee E, Kleber RJ, Jongmans MJ. Relational Patterns Between Caregivers With PTSD and Their Nonexposed Children: A Review. Trauma Violence Abuse. 2016 Apr;17(2):186-203. doi: 10.1177/1524838015584355. Epub 2015 May 11. PMID 25964276
- [Background] Wang Y, Chung MC, Wang N, Yu X, Kenardy J. Social support and posttraumatic stress disorder: A meta-analysis of longitudinal studies. Clin Psychol Rev. 2021 Apr;85:101998. doi: 10.1016/j.cpr.2021.101998. Epub 2021 Mar 4. PMID 33714168
- [Derived] Meijer L, Finkenauer C, Blankers M, de Gee A, Kramer J, Shields-Zeeman L, Thomaes K. Study protocol: development and randomized controlled trial of a preventive blended care parenting intervention for parents with PTSD. BMC Psychiatry. 2023 Feb 10;23(1):102. doi: 10.1186/s12888-023-04548-8. PMID 36765312